CLINICAL TRIAL: NCT06391372
Title: Effect of Local Estriol Treatment Before Vaginal Repair Surgery on Vaginal Tissues and Early Postoperative Pelvic Floor Functions
Brief Title: Effect of Local Estriol Treatment Before Vaginal Repair Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hatice Tukenmez Kurnaz (Other)
Responsible Party: Sponsor-Investigator, Hatice Tukenmez Kurnaz, Resident,M.D., Ankara University
Organization: Ankara University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023000504-2
Record Dates: First submitted 2024-04-05; First posted 2024-04-30 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Organ Prolapse; Pelvic Floor Disorders; Menopause; Vaginal Atrophy
Keywords: local estriol; colporrhaphy
MeSH Terms: conditions — Pelvic Organ Prolapse; Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: Patients who will be administered 1 g of intravaginal estriol via an applicator twice a week before going to bed for 4 preoperative weeks will constitute the study group. Patients who meet the same criteria as the study group and are not treated with local estriol will constitute the control group.
Who Masked: Outcomes Assessor
Masking Description: pathologist who will examine the tissue samples in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- local estriol (Experimental): Patients will receive 1 g of intravaginal estriol via an applicator twice a week before going to bed for 4 weeks preoperatively.
  Interventions: Drug: estriol cream
- control (No Intervention): Patients who met the same criteria as the study group and were not treated with local estriol

INTERVENTIONS:
Drug: estriol cream — 1 g intravaginal estriol via applicator twice a week before going to bed for 4 weeks
  Arms: local estriol

SUMMARY:
The aim of the study is to evaluate the effects of local estriol treatment applied before vaginal repair surgery on steroid receptors, inflammatory cell response, vascular, connective and nervous tissues in the vagina, and its effects on early postoperative period pelvic floor functions, satisfaction with the surgery and vaginal health.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is the herniation of pelvic organs into or beyond the vaginal walls and is a common health problem that affects daily activities and sexual function. Its negative impact on women's quality of life has been the subject of clinical research all over the world due to the economic burden it brings to the healthcare system.

The use of different classification systems for diagnosis and the fact that many women with mild prolapse are asymptomatic make it difficult to determine the exact prevalence of pelvic organ prolapse. Among women aged 50-79, the prevalence is 41% and the lifetime risk of prolapse surgery is 11%. This risk is expected to increase in the future.

Advancing age and postmenopausal status are known risk factors for pelvic organ prolapse. Since estradiol receptors alpha and beta (ESR1/2) are found in the squamous epithelium of the bladder, urethra, vagina, and pelvic floor muscles, it is evident that the pelvic organs and their surrounding muscle and connective tissue are sensitive to estrogen and that menopause is an important risk factor for the development of pelvic organ prolapse. The decline in estrogen during the postmenopausal period contributes not only to symptoms of pelvic organ prolapse but also to other pelvic floor disorders, including vulvovaginal atrophy, stress urinary incontinence (SUI), urge urinary incontinence (UUI), sexual dysfunction, and dyspareunia.

Studies show that estrogen levels have a significant impact on the function of the genital and lower urinary tract. Estrogen regulates the function of the vascular smooth muscles in the vaginal wall, affecting vaginal wall perfusion and smooth muscle tone. It also regulates bladder smooth muscle contractility, cellular and extracellular composition, and nerve density.

Local estrogen therapy (LET) works by increasing vaginal tissue blood flow, epithelial thickening, increased epithelial secretion and decrease in vaginal pH. From a physiological and psychosocial perspective, women using estrogen therapy describe positive effects such as normalization of sexual function, increased quality of life, improvement in relationships with their spouses, feeling 'less old', higher self-esteem and having a better social life.

In recent years, local estrogen therapy has become the focus of treatment of pelvic floor disorders. Various conservative and surgical methods have been described in the treatment of pelvic organ prolapse. Conservative treatment methods include topical estrogen. Among the surgical approaches, many vaginal and abdominal methods with or without graft material have been described. Surgical methods are mostly preferred in treatment.

The primary goal of POP surgery is to reduce symptoms and improve health-related quality of life. However, despite the continuous evolution in current surgical techniques, recurrence of symptoms is common. It is important to find ways to improve pelvic organ prolapse surgery outcomes. It is unclear whether preoperative LET is beneficial. Ismail and colleagues concluded in a Cochrane systematic review that further studies with long-term follow-up are needed to evaluate the effects of estrogen preparations before prolapse surgery.

The aim of this study is to evaluate the effects of preoperative local estriol application on the vaginal tissues and the effects of preoperative local estriol application on early postoperative period pelvic floor functions, satisfaction with the surgery and vaginal health in postmenopausal women planned for vaginal repair surgery.

As a result, steroid receptors (ER, PR, AR), immune cell types and distribution, CD34 and vascular endothelial density, collagen fiber density, S100 in the anterior and/or posterior vaginal wall in patients with and without local estriol treatment before colporrhaphy anterior and/or posterior. The difference in nerve fiber density and epithelial maturation index levels will be investigated. In addition, the Pelvic Floor Distress Inventory (PFDI-20), which is valid in Turkish, Pelvic Floor Impact Questionnaire (PFIQ-7), Patient General Impression of Improvement (PGI-I) and VAS scoring and early postoperative pelvic floor functions were evaluated in the study and control groups before and after surgery. and patient satisfaction regarding the surgery will be compared. There will also be comparisons between the pre-surgical study and control group through the vaginal health index (VHI), which is a quantitative assessment of vaginal health. Follow-ups are planned to be carried out with the patients' routine check-up visits to the hospital.

ELIGIBILITY:
Inclusion Criteria:

-Postmenopausal women with a diagnosis of pelvic organ prolapse and an indication for vaginal repair surgery including colporrhaphy anterior and/or posterior surgery

Exclusion Criteria:

* Psychiatric and neurological disease that causes disability in mental and motor functions
* receiving systemic/local hormone replacement therapy in the last three months
* applying vulvar/local steroids for any reason within the last three months
* receiving treatment for pelvic and/or lower genital tract infection in the last three months
* history of malignancy
* previous vaginal repair surgery with/without mesh

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Morphological examinations of vaginal tissues obtained after surgery from the study and control groups | 4 weeks after starting local estriol treatment
  1x0.5 cm tissue samples, made by Ankara University Faculty of Medicine, Department of Medical Pathology, will be taken from the vaginal tissues obtained after surgery from the study and control groups. After paraffin blocking, Epithelial thickness will be evaluated during routine histopathological evaluation with H.E staining. Epithelial thickness will be evaluated in micrometers
Immunohistochemical examinations of vaginal tissues obtained after surgery from the study and control groups | 4 weeks after starting local estriol treatment
  Sections obtained from the blocks will be sectioned with 6 samples per glass, and steroid receptors (ER, PR, AR), CD3/CD20/CD68/CD4/CD8, CD34 and S100 will be stained with the Ventana automatic staining device and as secondary antibodies. (A total of 60 immunohistochemical tests will be performed in 6 glasses of 10 antibodies to be studied). With these dyes, the presence and density of CD3/CD20/CD68/CD4/CD8 and inflammatory cells in the epithelial and subepithelial tissue and the type distribution of immune cells will be determined. Vascular endothelial density will be evaluated with CD34 and nerve fiber density will be evaluated with S100.
Morphological examinations of vaginal tissues obtained after surgery from the study and control groups | 4 weeks after starting local estriol treatment
  The alignment and maturation of vaginal epithelial squamous cells will be evaluated during routine histopathological evaluation. Alignment and maturation of squamous cells will be evaluated as a percentage.
Morphological examinations of vaginal tissues obtained after surgery from the study and control groups | 4 weeks after starting local estriol treatment
  Connective tissue changes in the vaginal subepithelial area will be evaluated during routine histopathological evaluation. Connective tissue change in the subepithelial area will be evaluated as a percentage.
Morphological examinations of vaginal tissues obtained after surgery from the study and control groups | 4 weeks after starting local estriol treatment
  Distribution of vaginal vascular structures will be evaluated during routine histopathological evaluation. Distribution of vascular structures will be evaluated as a percentage.

SECONDARY OUTCOMES:
Turkish version of Pelvic Floor Distress Inventory-20 (PFDI-20) was used to evaluate pelvic floor functions in the study and control groups. | The determined questionnaires will be administered to the patients 4 weeks before the surgical procedure, before the surgery and 4 weeks after the surgery.
  The PFDI-20 Scale includes 20 items with 3 subscales:POPDI-6,UDI-6, and CRADI-8. The total score of the scale is between 0-300. The best score that can be obtained from the entire survey is 0, the worst score is 300. The higher the score obtained as a result of this survey, the greater the degree of complaint of pelvic floor dysfunction.
Patient Global Improvement Impression Scale (PGI-I) was used to understand the change in the patient's complaints after vaginal repair surgery in the treatment and control groups. | 4 weeks after surgery
  The Patient Global Impression of Improvement Scale (PGI-I) is a tool designed to measure patient interpretation of symptom changes following intervention. We will use it in this study to understand the change in the patient's complaints after vaginal repair surgery in the treatment and control groups. In this way, we will avoid relying on disease-specific questions and the inherent researcher bias that may be present in these questions. PGI-I score was recorded on a 7-point scale where 1 = very much better/improved, 2 = much better/improved, 3 = a little better/improved, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse.
Questioning the feeling of pain/discomfort in the vagina after surgery using VAS | 4 weeks after surgery
  Questioning the feeling of pain/discomfort in the vagina after surgery using VAS; We aim to compare the effect of local estriol treatment applied in the preoperative period on these complaints.
To evaluate the effect of preoperative local estirol treatment on vaginal health in the preoperative period between the study and control groups using the vaginal health index (VHI). | 4 weeks before and before surgery
  Vaginal health index (VHI), a quantitative assessment of vaginal health, is used to evaluate vaginal elasticity, fluid volume, vaginal pH level, epithelial integrity, and changes in moisture. The VHI scale is interpreted as ranging from 5 points (severe) to 25 points (normal) on all five parameters. The vaginal health index will be determined in line with the vaginal examination performed by me 4 weeks before and just before the operation. In this way, the effect of preoperative local estirol treatment on vaginal health in the preoperative period will be compared between the study and control groups.
Turkish version of Pelvic Floor Impact Questionnaire (PFIQ-7) was used to evaluate pelvic floor functions in the study and control groups. | Determined questionnaires will be administered to patients 4 weeks before the surgical procedure, before surgery, and 4 weeks after the surgery.
  The Pelvic Floor Impact Questionnaire (PFIQ-7) is a functional status measure that assesses the degree of impact of a person's bowel, bladder, and/or pelvic symptoms on different activities of daily living, social relationships, or emotions. It also has three scales: POPIQ-7; UIO-7; and CRAIQ-7. In the form, patients' complaints were none (0); less (1); middle (2); many (3); It is rated as.
  Total score ranges from 0 to 21. Lower score means less quality of life impact expresses.
VAS scoring for postmenopausal genitourinary syndrome complaints in the study and control groups | Determined questionnaires will be administered to patients 4 weeks before the surgical procedure, before surgery, and 4 weeks after the surgery.
  Through VAS evaluation, the severity of genital burning, genital dryness, genital itching and dysuria symptoms of the patients in the study and control groups will be scored between 0-10. Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically into numerical values.No complaints are scored as 0 points and complaints of the worst severity imaginable are rated as 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Dokmeci, Study Director — Ankara University Faculty of Medicine, Department of Gynecology and Obstetrics
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maher C, Feiner B, Baessler K, Schmid C. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD004014. doi: 10.1002/14651858.CD004014.pub5. PMID 23633316
- [Background] Wu JM, Matthews CA, Conover MM, Pate V, Jonsson Funk M. Lifetime risk of stress urinary incontinence or pelvic organ prolapse surgery. Obstet Gynecol. 2014 Jun;123(6):1201-1206. doi: 10.1097/AOG.0000000000000286. PMID 24807341
- [Background] Wu JM, Vaughan CP, Goode PS, Redden DT, Burgio KL, Richter HE, Markland AD. Prevalence and trends of symptomatic pelvic floor disorders in U.S. women. Obstet Gynecol. 2014 Jan;123(1):141-148. doi: 10.1097/AOG.0000000000000057. PMID 24463674
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Lang JH, Zhu L, Sun ZJ, Chen J. Estrogen levels and estrogen receptors in patients with stress urinary incontinence and pelvic organ prolapse. Int J Gynaecol Obstet. 2003 Jan;80(1):35-9. doi: 10.1016/s0020-7292(02)00232-1. PMID 12527458
- [Background] Weber MA, Limpens J, Roovers JP. Assessment of vaginal atrophy: a review. Int Urogynecol J. 2015 Jan;26(1):15-28. doi: 10.1007/s00192-014-2464-0. Epub 2014 Jul 22. PMID 25047897
- [Background] Kim NN, Min K, Pessina MA, Munarriz R, Goldstein I, Traish AM. Effects of ovariectomy and steroid hormones on vaginal smooth muscle contractility. Int J Impot Res. 2004 Feb;16(1):43-50. doi: 10.1038/sj.ijir.3901138. PMID 14963470
- [Background] Kim SW, Kim NN, Jeong SJ, Munarriz R, Goldstein I, Traish AM. Modulation of rat vaginal blood flow and estrogen receptor by estradiol. J Urol. 2004 Oct;172(4 Pt 1):1538-43. doi: 10.1097/01.ju.0000137744.12814.2e. PMID 15371887
- [Background] Ibe C, Simon JA. Vulvovaginal atrophy: current and future therapies (CME). J Sex Med. 2010 Mar;7(3):1042-50; quiz 1051. doi: 10.1111/j.1743-6109.2009.01692.x. PMID 20500443
- [Background] Rahn DD, Ward RM, Sanses TV, Carberry C, Mamik MM, Meriwether KV, Olivera CK, Abed H, Balk EM, Murphy M; Society of Gynecologic Surgeons Systematic Review Group. Vaginal estrogen use in postmenopausal women with pelvic floor disorders: systematic review and practice guidelines. Int Urogynecol J. 2015 Jan;26(1):3-13. doi: 10.1007/s00192-014-2554-z. Epub 2014 Nov 13. PMID 25392183
- [Background] Weber MA, Kleijn MH, Langendam M, Limpens J, Heineman MJ, Roovers JP. Local Oestrogen for Pelvic Floor Disorders: A Systematic Review. PLoS One. 2015 Sep 18;10(9):e0136265. doi: 10.1371/journal.pone.0136265. eCollection 2015. PMID 26383760
- [Background] Raju R, Linder BJ. Evaluation and Management of Pelvic Organ Prolapse. Mayo Clin Proc. 2021 Dec;96(12):3122-3129. doi: 10.1016/j.mayocp.2021.09.005. PMID 34863399
- [Background] Barber MD, Brubaker L, Nygaard I, Wheeler TL 2nd, Schaffer J, Chen Z, Spino C; Pelvic Floor Disorders Network. Defining success after surgery for pelvic organ prolapse. Obstet Gynecol. 2009 Sep;114(3):600-609. doi: 10.1097/AOG.0b013e3181b2b1ae. PMID 19701041
- [Background] Diwadkar GB, Barber MD, Feiner B, Maher C, Jelovsek JE. Complication and reoperation rates after apical vaginal prolapse surgical repair: a systematic review. Obstet Gynecol. 2009 Feb;113(2 Pt 1):367-73. doi: 10.1097/AOG.0b013e318195888d. PMID 19155908
- [Background] Ismail SI, Bain C, Hagen S. Oestrogens for treatment or prevention of pelvic organ prolapse in postmenopausal women. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD007063. doi: 10.1002/14651858.CD007063.pub2. PMID 20824855
- [Background] Kaplan PB, Sut N, Sut HK. Validation, cultural adaptation and responsiveness of two pelvic-floor-specific quality-of-life questionnaires, PFDI-20 and PFIQ-7, in a Turkish population. Eur J Obstet Gynecol Reprod Biol. 2012 Jun;162(2):229-33. doi: 10.1016/j.ejogrb.2012.03.004. Epub 2012 Apr 4. PMID 22480412
- [Background] Hossack T, Woo H. Validation of a patient reported outcome questionnaire for assessing success of endoscopic prostatectomy. Prostate Int. 2014 Dec;2(4):182-7. doi: 10.12954/PI.14066. Epub 2014 Dec 30. PMID 25599074
- [Background] Samuels JB, Garcia MA. Treatment to External Labia and Vaginal Canal With CO2 Laser for Symptoms of Vulvovaginal Atrophy in Postmenopausal Women. Aesthet Surg J. 2019 Jan 1;39(1):83-93. doi: 10.1093/asj/sjy087. PMID 29726916